CLINICAL TRIAL: NCT03274726
Title: Iron Status of Toddlers, Non-pregnant, and Pregnant Women in the United States
Brief Title: Iron Status of Women and Young Children in the United States
Acronym: NHANES
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Priya Gupta, ORISE Fellow, Centers for Disease Control and Prevention
Other Study IDs: CDC-NCCDPHP-2011-17
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Iron-deficiency; Nutritional Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency; Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This analysis describes the distribution of TBI and the prevalence of iron deficiency (ID) and iron deficiency anemia (IDA) among toddlers, non-pregnant women, and pregnant women.

DETAILED DESCRIPTION:
Background: Total body iron stores (TBI), which are calculated from serum ferritin (SF) and soluble transferrin receptor (sTfR) concentrations, can be used to assess the iron status of populations in the United States.

Objective: This analysis describes the distribution of TBI and the prevalence of iron deficiency (ID) and iron deficiency anemia (IDA) among toddlers, non-pregnant women, and pregnant women.

Design: Investigators analyzed data from NHANES; toddlers aged 12-23 mo (NHANES 2003-2010), non-pregnant women aged 15-49 y (NHANES 2007-2010), and pregnant women aged 12-49 y (NHANES 1999-2010). Investigators used SAS survey procedures to plot distributions of TBI and produce prevalence estimates of ID and IDA for each target population. All analyses were weighted to account for the complex survey design

ELIGIBILITY:
Included:

* Children ages 12-23 months and Women ages 12-49 years
* Those who completed the MEC

Excluded:

- Those missing data on iron biomarkers

Ages: 12 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: NHANES is a nationally-representative, cross-sectional study of nutrition and health for individuals residing in the U.S.
Sampling Method: Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2010-12-01 (Actual); Study Completion 2010-12-01 (Actual)

PRIMARY OUTCOMES:
Iron Deficiency | 1999-2010
  Total Body Iron <0 mg/kg

REFERENCES:
- [Derived] Gupta PM, Hamner HC, Suchdev PS, Flores-Ayala R, Mei Z. Iron status of toddlers, nonpregnant females, and pregnant females in the United States. Am J Clin Nutr. 2017 Dec;106(Suppl 6):1640S-1646S. doi: 10.3945/ajcn.117.155978. Epub 2017 Oct 25. PMID 29070559